CLINICAL TRIAL: NCT04760431
Title: Anti-HER2 TKI Versus Pertuzumab in Combination With Dose-dense Trastuzumab and Taxane as First Line in HER2-positive Breast Cancer Patients With Active Brain Metastases: A Phase II, Multicenter, Double-blind, Randomized Clinical Trial
Brief Title: TKIs vs. Pertuzumab in HER2+ Breast Cancer Patients With Active Brain Metastases (HER2BRAIN)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Peking University International Hospital (Other); Sun Yat-sen University (Other); Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HER2BRAIN
Record Dates: First submitted 2021-01-25; First posted 2021-02-18 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-01

CONDITIONS: HER2-positive Breast Cancer; Brain Metastases
Keywords: HER2-positive Breast Cancer; Brain Metastases; Tyrosine kinase inhibitors
MeSH Terms: conditions — Brain Neoplasms | interventions — Trastuzumab; Taxoids; Docetaxel; Paclitaxel; pertuzumab; Tyrosine Kinase Inhibitors; pyrotinib; neratinib; tucatinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Trastuzumab, Taxanes and Pertuzumab
  Interventions: Drug: Trastuzumab; Drug: Taxanes; Drug: Pertuzumab
- Group B (Experimental): Trastuzumab, Taxanes and TKIs
  Interventions: Drug: Trastuzumab; Drug: Taxanes; Drug: Tyrosine kinase inhibitor

INTERVENTIONS:
Drug: Trastuzumab — 8 mg/kg loading dose for Cycle 1, followed by 6 mg/kg for subsequent cycles, administered by IV infusion every week until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Herceptin
Drug: Taxanes — Docetaxel: 75 mg/m2, administered by IV infusion every 3 weeks Paclitaxel: 175 mg/m2, administered by IV infusion every 3 weeks Paclitaxel (Albumin bound): 260 mg/m2, administered by IV infusion every 3 weeks Paclitaxel Liposome: 135-175 mg/m2, administered by IV infusion every 3 weeks
  Other Names: Docetaxel, Paclitaxel, Paclitaxel (Albumin bound), Paclitaxel Liposome
Drug: Pertuzumab — 840 milligrams (mg) loading dose of pertuzumab, followed every 3 weeks thereafter by a dose of 420 mg via intravenous (IV) infusion until disease progression, unacceptable toxicity, withdrawal of consent, or study termination.
  Other Names: Perjeta
  Arms: Group A
Drug: Tyrosine kinase inhibitor — Pyrotinib: 400mg po within 30 minutes after a meal, QD, every 3 weeks Neratinib: 240mg po QD, every 3 weeks Tucatinib: 300mg po Q12H
  Other Names: Pyrotinib, Neratinib, Tucatinib
  Arms: Group B

SUMMARY:
This is a prospective, randomized, 2-arm, Phrase 2, superiority and multicenter study to compare the efficiency of Anti-HER2 TKI versus Pertuzumab in Combination With Dose-dense Trastuzumab and Taxane in HER2-positive breast cancer patients with active refractory brain metastases.

DETAILED DESCRIPTION:
This is a prospective, randomized, 2-arm, Phrase 2, superiority and multicenter study. HER2-positive breast cancer patients with active refractory brain metastases are included. There will be two group: Group A (Trastuzumab, Taxanes and Pertuzumab) and Group B (Trastuzumab, Taxanes and TKIs). The primary outcome is objective response rate (ORR).

ELIGIBILITY:
Inclusion Criteria:

1. Patients provided written informed consent
2. Women aged 18-75 years
3. Histologically or cytologically confirmed HER2-positive (IHC 3+ or ISH+) breast cancer
4. Patients of HER2 positive breast cancer with a documented central nervous system (CNS) recurrence/progression (by imaging) during or after Trastuzumab based therapy
5. At least one measurable and progressive lesion in the CNS (≥10 mm on T1-weighted, gadolinium-enhanced MRI)
6. Previous treatment with HER2 inhibitors to be discontinued prior to first study treatment administration (at least 14 days for trastuzumab and other antibodies, at least 7 days for lapatinib)
7. Previous chemotherapy and hormonal therapy (adjuvant and metastatic regimens) allowed, but chemotherapy must have been discontinued at least 14 days and hormonal therapy at least 7 days prior to first study treatment administration
8. Prior surgery, whole brain radiotherapy or stereotactic radiosurgery allowed provided that there is unequivocal evidence of one or more new and/or progressive brain metastases after completion of whole brain radiotherapy or stereotactic radiosurgery
9. Previous radiotherapy allowed, but radiotherapy must have been discontinued at least 14 days prior to first study treatment administration
10. Normal cardiac function
11. Patients must have recovered to baseline condition or to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade = 1 from any acute CTCAE v. 5.0 grade =2 side effects of previous treatments
12. Without infection of human immunodeficiency virus (HIV) on central laboratory assay results prior to randomization
13. Alanine aminotransferase (ALT) </= 2.5 × the upper limit of normal (ULN), Aspartate aminotransferase (AST) </= 2.5 × ULN prior to randomization
14. Total bilirubin (TBIL) </= 1.25 × ULN
15. Alkaline phosphatase (ALK) </= 2.5 × ULN
16. Gamma glutamyl transpeptidase (GGT) </= 2.5 × ULN
17. Albumin >/= 30g/L
18. Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1
19. A life expectancy of at least 1 month
20. Women of child-bearing age should take effective contraceptive measures
21. Serum total bilirubin (TBil) </= 1.5 × ULN
22. Serum creatinine (Scr) </= 1.5 × ULN
23. WBC >/= 3×109/L, Blood neutrophil count >/= 1×109/L, Platelet count >/= 100×109/L, HB >/= 9 g/dL

Exclusion Criteria:

1. Lack of histological or cytological confirmation of HER2-positive (IHC 3+ or ISH-positive) breast cancer
2. Cerebral hernia
3. Need radiotherapy or surgery immediately
4. Active cerebral infarction or hemorrhage
5. Only meningeal metastasis
6. Earlier exposure to doxorubicin or pirarubicin at a dosage of more than 360 mg/m2
7. Earlier exposure to epirubicin at a dosage of more than 900 mg/m2
8. Prior treatment with HER2-tyrosine kinase inhibitors
9. Treatment with trastuzumab emtansine within 6 months
10. Any other current malignancy or malignancy diagnosed within the past five years (other than carcinoma in situ or stage Ia carcinoma of the cervix, skin basal cell carcinoma and papillary thyroid carcinoma at early stage)
11. Active infection with human immunodeficiency virus (HIV) prior to first study treatment administration.
12. History of participating any other clinical trials within 30 days prior to randomization
13. Known hypersensitivity (Grade 3 or 4) to any of the trial drugs
14. Pregnancy or lactation
15. Current severe systemic disease (for example, clinically significant cardiovascular, pulmonary, or renal disease)
16. Legal incompetence or limitation.
17. Considered unable to complete the study or sign the informed consent due to a medical or mental disorder by the investigator.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | up to 3 years
  The sum of complete response (CR) rate and partial response (PR) rate by measurement of target lesions (intracranial lesions)

SECONDARY OUTCOMES:
Objective Response Rate 2 (ORR2) | up to 3 years
  The sum of complete response (CR) rate and partial response (PR) rate by measurement of extracranial lesions
Progression-free Survival (PFS) | up to 3 years
  PFS is defined as time from randomization to disease progression or death, whichever occurs first.
  Progression of disease was determined if at least 1 of the following criteria applied:
  1. At least a 20% increase in the sum of the diameters (SoD) of target lesions taking as reference the smallest SoD recorded since the treatment started, together with an absolute increase in the SoD of at least 5 mm
  2. Appearance of 1 or more new lesions
  3. Unequivocal progression of existing non-target lesions
Overall Survival (OS) | up to 3 years
  OS is defined as time from randomization to death for any cause. If there is no death reported for a subject before the date cutoff for OS analysis, OS will be censored at the last contact date at which the subject is known to be alive.
  For patients who had not died up to the cut-off date, the date they were last known to be alive was derived from the patient status records, the trial completion record, radiological imaging assessments, the study treatment termination record, and the randomization date.
Clinical benefit rate (CBR) | up to 3 years
  CBR is defined as the sum of CR rate, PR rate, and more than 6 months' SD (stable disease) rate
Disease control rate (DCR) | up to 3 years
  DCR is defined that the sum of CR rate, PR rate, and SD rate.
Peripheral neurotoxicity | 30 days after last treatment
  Peripheral neurotoxicities are defined as the number of patients who suffer from neurotoxicities (NCI CTCAE v5.0)

CONTACTS AND LOCATIONS:
Overall Officials: Xuexin He, MD, Principal Investigator — Second Affiliated Hospital, Zhejiang University, School of Medicine
Locations (3):
- China (3):
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - First Affiliated Hospital, Zhejiang University, School of Medicine, Hangzhou, Zhejiang